CLINICAL TRIAL: NCT00824083
Title: Functional and Clinical Long-Term Outcome of Ewing Sarcoma Treatment
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01ER0807
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Sarcoma, Ewing's
Keywords: bone tumors; long-term function; daily activity; late sequelae
MeSH Terms: conditions — Sarcoma, Ewing; Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: sarcoma survivors
- 2: healthy subjects

SUMMARY:
The purpose of the study is to assess the functional outcome, quality of life and late sequelae in a representative sample of 600 long-term survivors of Ewing sarcoma and to build a unique clinical and functional data pool of the underlying cohort of 3000 Ewing sarcoma patients with a follow-up of 3 decades.

DETAILED DESCRIPTION:
Trial objective: As survival rates of bone sarcoma patients have been raised owing to improved treatment strategies the focus of investigations is now on the medical, social, and economic sequelae of intensive multimodal treatment. This study aims to assess the functional outcome, quality of life and late sequelae in a representative sample of long-term survivors of Ewing sarcoma. The data recorded combined with standardized treatment data covering a 30-year period will produce a data pool that is unique for its magnitude and will be used for the development of guidelines for further improvements of future bone sarcoma treatment.

Working plan: The working plan provides for the assessment of functional outcome and quality of life by means of validated tools (TESS, SF36, PEDQOL) and objectively measuring daily activity patterns by using the Step Activity Monitor (SAM) in 600 long-term Ewing sarcoma survivors and a control group of 300 matched healthy subjects. Information on sarcoma treatment and follow-up is obtained by re-structuring and complementing the database of the relevant patient cohort (n=3000) from four consecutive nationwide and international clinical trials between 1980 and 2008. Procedures of local treatment will be evaluated regarding functional outcome, quality of life, and survival probability and prognostic factors predicting long-term outcome will be identified.

Exploitation of results: The results will be presented at scientific meetings and will be published in international journals. Guidelines will be developed regarding improvements in the treatment, rehabilitation, and social integration of bone sarcoma patients to be utilized in guiding patients and in the decision process of medical professionals regarding their treatment. In the long run, the evidence based guidelines on treatment and follow-up are to be transferred into the health system.

ELIGIBILITY:
Inclusion Criteria:

* CESS81/CESS86/EICESS92/EURO-E.W.I.N.G.99 trials participants of the German Society of Pediatric Hematology and Oncology (GPOH)

Exclusion Criteria:

* no complete remission (CR)
* any kind of paralysis
* <3y after diagnosis

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Ewing sarcoma survivors and 1:2 matched control group of healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2009-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
physical activity (SAM: step-activity-monitor) | 3-30years after primary diagnosis of Ewing sarcoma

SECONDARY OUTCOMES:
health-related quality of life (SF36, PEDQOL) | 3-30years after primary diagnosis of Ewing sarcoma
functional status (TESS) | 3-30years after primary diagnosis of Ewing sarcoma
psychological status (HADS, BIS-BAS) | 3-30years after primary diagnosis of Ewing sarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ranft, Dr., Principal Investigator — University Hospital Muenster; Heribert Jürgens, Prof., Study Chair — University Hospital Muenster
Locations (2):
- Germany (2):
  - Department of Pediatric Hematology and Oncology, University Children's Hospital, Münster, North Rhine-Westphalia
  - Motion Analysis Lab, Orthopedic Department, University Hospital, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandes M, Schomaker R, Mollenhoff G, Rosenbaum D. Quantity versus quality of gait and quality of life in patients with osteoarthritis. Gait Posture. 2008 Jul;28(1):74-9. doi: 10.1016/j.gaitpost.2007.10.004. Epub 2007 Nov 28. PMID 18054233
- [Background] Gerber LH, Hoffman K, Chaudhry U, Augustine E, Parks R, Bernad M, Mackall C, Steinberg S, Mansky P. Functional outcomes and life satisfaction in long-term survivors of pediatric sarcomas. Arch Phys Med Rehabil. 2006 Dec;87(12):1611-7. doi: 10.1016/j.apmr.2006.08.341. PMID 17141641
- [Background] Hoffmann C, Gosheger G, Gebert C, Jurgens H, Winkelmann W. Functional results and quality of life after treatment of pelvic sarcomas involving the acetabulum. J Bone Joint Surg Am. 2006 Mar;88(3):575-82. doi: 10.2106/JBJS.D.02488. PMID 16510825
- [Background] McDonald CM, Widman L, Abresch RT, Walsh SA, Walsh DD. Utility of a step activity monitor for the measurement of daily ambulatory activity in children. Arch Phys Med Rehabil. 2005 Apr;86(4):793-801. doi: 10.1016/j.apmr.2004.10.011. PMID 15827934
- [Background] Nagarajan R, Neglia JP, Clohisy DR, Robison LL. Limb salvage and amputation in survivors of pediatric lower-extremity bone tumors: what are the long-term implications? J Clin Oncol. 2002 Nov 15;20(22):4493-501. doi: 10.1200/JCO.2002.09.006. PMID 12431974
- [Background] Paulussen M, Craft AW, Lewis I, Hackshaw A, Douglas C, Dunst J, Schuck A, Winkelmann W, Kohler G, Poremba C, Zoubek A, Ladenstein R, van den Berg H, Hunold A, Cassoni A, Spooner D, Grimer R, Whelan J, McTiernan A, Jurgens H; European Intergroup Cooperative Ewing's Sarcoma Study-92. Results of the EICESS-92 Study: two randomized trials of Ewing's sarcoma treatment--cyclophosphamide compared with ifosfamide in standard-risk patients and assessment of benefit of etoposide added to standard treatment in high-risk patients. J Clin Oncol. 2008 Sep 20;26(27):4385-93. doi: 10.1200/JCO.2008.16.5720. PMID 18802150
- [Background] Pieper S, Ranft A, Braun-Munzinger G, Jurgens H, Paulussen M, Dirksen U. Ewing's tumors over the age of 40: a retrospective analysis of 47 patients treated according to the International Clinical Trials EICESS 92 and EURO-E.W.I.N.G. 99. Onkologie. 2008 Dec;31(12):657-63. doi: 10.1159/000165361. Epub 2008 Nov 20. PMID 19060503
- [Background] Rodl RW, Hoffmann C, Gosheger G, Leidinger B, Jurgens H, Winkelmann W. Ewing's sarcoma of the pelvis: combined surgery and radiotherapy treatment. J Surg Oncol. 2003 Jul;83(3):154-60. doi: 10.1002/jso.10256. PMID 12827683
- [Background] Rosenbaum D, Brandes M, Hardes J, Gosheger G, Rodl R. Physical activity levels after limb salvage surgery are not related to clinical scores-objective activity assessment in 22 patients after malignant bone tumor treatment with modular prostheses. J Surg Oncol. 2008 Aug 1;98(2):97-100. doi: 10.1002/jso.21091. PMID 18521841
- [Background] Schuck A, Ahrens S, Paulussen M, Kuhlen M, Konemann S, Rube C, Winkelmann W, Kotz R, Dunst J, Willich N, Jurgens H. Local therapy in localized Ewing tumors: results of 1058 patients treated in the CESS 81, CESS 86, and EICESS 92 trials. Int J Radiat Oncol Biol Phys. 2003 Jan 1;55(1):168-77. doi: 10.1016/s0360-3016(02)03797-5. PMID 12504050
- [Background] Song KM, Bjornson KF, Cappello T, Coleman K. Use of the StepWatch activity monitor for characterization of normal activity levels of children. J Pediatr Orthop. 2006 Mar-Apr;26(2):245-9. doi: 10.1097/01.bpo.0000218532.66856.6c. PMID 16557143
- [Background] Weddington WW. Psychological outcomes in survivors of extremity sarcomas following amputation or limb-sparing surgery. Cancer Treat Res. 1991;56:53-60. doi: 10.1007/978-1-4615-3896-7_5. No abstract available. PMID 1681879